CLINICAL TRIAL: NCT05521438
Title: A Multicenter, Randomized, Vehicle-Controlled, Double-Blind, Parallel Comparison Study of QRX003 Lotion in Subjects With Netherton Syndrome
Brief Title: Safety, Tolerability and Efficacy of QRX003 Lotion in Subjects With Netherton Syndrome
Status: Active, not recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Quoin Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CL-QRX003-001
Record Dates: First submitted 2022-08-17; First posted 2022-08-30 (Actual); Last update posted 2025-10-28 (Actual); Status verified 2025-03

CONDITIONS: Netherton Syndrome
MeSH Terms: conditions — Netherton Syndrome

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Masking Description: Double-blind
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- QRX003-2% QAM (Experimental): Subjects will apply test article once daily in the morning (QAM) for 12 weeks
  Interventions: Drug: QRX003-2% Lotion
- QRX003-4% QAM (Experimental): Subjects will apply test article once daily in the morning (QAM) for 12 weeks
  Interventions: Drug: QRX003-4% Lotion QAM
- Vehicle Lotion (Experimental): Subjects will apply test article once daily in the morning (QAM) for 12 weeks
  Interventions: Drug: Vehicle
- QRX003-4% BID (Experimental): Subjects will apply test article twice daily BID for 12 weeks
  Interventions: Drug: QRX003-4% Lotion BID

INTERVENTIONS:
Drug: QRX003-2% Lotion — QRX003Topical Lotion containing 2% active drug (serine protease inhibitor)
  Arms: QRX003-2% QAM
Drug: QRX003-4% Lotion QAM — QRX003Topical Lotion containing 4% active drug (serine protease inhibitor)
  Arms: QRX003-4% QAM
Drug: Vehicle — Vehicle Lotion
  Arms: Vehicle Lotion
Drug: QRX003-4% Lotion BID — QRX003Topical Lotion containing 4% active drug (serine protease inhibitor)
  Arms: QRX003-4% BID

SUMMARY:
This study has been designed to determine the safety, tolerability and efficacy of QRX003 lotion 2%, 4% QAM or 4% BID in subjects with Netherton Syndrome (NS) in comparison to vehicle

ELIGIBILITY:
Inclusion Criteria:

* Subject is a male or non-pregnant female at least 14 years of age.
* Females must be post-menopausal , surgically sterile , or use an effective method of birth control , for the duration of the study and for 3 months following completion of treatment. Women of childbearing potential (WOCBP) must have a negative urine pregnancy test (UPT) at Visit 1/Screening and Visit 2/Baseline.
* Subject has a clinical diagnosis of NS and agrees to genetic testing at Visit 1/Screening for confirmation of NS diagnosis if the subject does not have test results confirming a SPINK5 mutation.
* Subject has NS lesions in the Treatment Area (i.e., arms or lower legs).
* Subject is in good general health and free of any disease state or physical condition that might impair evaluation of NS or exposes the subject to an unacceptable risk by study participation.

Exclusion Criteria:

* Subject is pregnant, lactating, or is planning to become pregnant during the study.
* Subject has any skin pathology in the Treatment Area or condition that, could interfere with the evaluation of the test article or requires use of interfering topical, systemic, or surgical therapy.
* Subject has Fridericia-corrected QT ≥ 450 ms for males or ≥ 470 ms for females
* Subject has active cancer of any type excluding non-melanoma skin cancer outside of the Treatment Area.
* Subject has diabetes of any type, except non-insulin dependent diabetes mellitus that is reasonably controlled.
* Subject has evidence of active infection during screening, or serious infection within 30 days prior to Visit 2/Baseline.
* Subject has known human immunodeficiency virus, hepatitis B or C virus, or active or latent tuberculosis.
* Subject has used ultraviolet phototherapy within the Treatment Area within 4 weeks prior to Visit 2/Baseline.
* Subject has used systemic prescription treatment for NS within 4 weeks prior to Visit 2/Baseline.
* Subject has used systemic biologic therapy for NS.
* Subject has used topical prescription treatment in the Treatment Area within 2 weeks prior to Visit 2/Baseline.
* Subject has used any topical bland moisturizers/emollients in the Treatment Area within 24 hours prior to Visit 2/Baseline.
* Subject is currently enrolled in an investigational drug, biologic, or device study.
* Subject has used an investigational drug, biologic, or device treatment within 30 days prior to Visit 2/Baseline.

Min Age: 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-06-23 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Efficacy Endpoints-1-point IGA | Up to week 16
  Proportion of subjects with 1-point reduction on the Investigator's Global Assessment (IGA) from Baseline. The IGA assesses overall severity of a subject's NS based on a 5-point scale where 0 = clear, 1 = almost clear, 2 = mild, 3 = moderate, and 4 = severe.
Efficacy Endpoints-2-point IGA | Up to week 16
  Proportion of subjects with 2-point reduction in IGA from Baseline.
Efficacy Endpoints-NS Sign | Up to week 16
  Change from Baseline in each individual NS Sign (erythema and scaling). Severity of each NS sign is graded on a 5-point scale.
Efficacy Endpoints-BSA | Up to week 16
  Change from Baseline in total Body Surface Area (BSA) affected by NS in the Treatment Area
Efficacy Endpoints-WI-NRS score | Up to week 16
  Change from Baseline in the Worst Itch-Numeric Rating Scale (WI-NRS) score. Itch severity is graded on an 11-point scale where 0 represents "no itch" and 10 represents "worst itch imaginable".
Efficacy Endpoints-TSQM | Up to week 16
  Assessment of subject satisfaction with treatment based on the Treatment Satisfaction Questionnaire for Medication (TSQM). The TSQM measures a subject's level of satisfaction or dissatisfaction with the treatment. Composite scores can range from 0 to 100; higher scores indicate better satisfaction.
Efficacy Endpoints-Rescue Therapy | Up to week 16
  Proportion of subjects requiring rescue therapy
Safety Endpoints-AEs | Up to week 16
  Any local and systemic AEs (Adverse Events)/serious AEs
Safety Endpoints-LSR | Up to week 16
  Number of subjects with presence of the following LSRs (Local Skin Reactions): edema, excoriations, oozing/vesiculation/crusting, and erosions at any study visit.

CONTACTS AND LOCATIONS:
Overall Officials: Tony Andrasfay, Study Director — Therapeutics, Inc.
Locations (5):
- United States (5):
  - Site #1, San Diego, California
  - Site #4, Indianapolis, Indiana
  - Site #5, Quincy, Massachusetts
  - Site #3, Charleston, South Carolina
  - Site #2, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: No